CLINICAL TRIAL: NCT07237529
Title: What is the Feasibility and Potential Impact of Narrative Exposure Therapy (NET) for People Experiencing Psychosis?
Brief Title: What is the Feasibility of Narrative Exposure Therapy (NET) for People Experiencing Psychosis?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25052
Record Dates: First submitted 2025-09-19; First posted 2025-11-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Psychosis; Schizophrenia and Other Psychotic Disorders
Keywords: Narrative Exposure Therapy; Psychosis; Trauma; Intervention Study
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a single group assignment. All participants will get the same intervention, Narrative Exposure Therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Exposure Therapy (NET) Arm (Experimental): In Narrative Exposure Therapy (NET), patients construct a detailed narration of their life story with the therapist, focusing on integrating traumatic memories into a coherent whole, including sensory, cognitive, emotional, and physiological aspects. The therapist documents the testimony. After an initial evaluation, including a questionnaire (TALE in this study), patients receive psychoeducation about trauma symptoms, followed by a preparatory introduction. Therapy begins with creating a "lifeline," an autobiographic overview of positive and traumatic events. Patients then undergo "Narrative Exposure," chronologically recounting their life story with in-depth exploration of emotionally charged experiences, particularly trauma, to contextualize and integrate them into reorganized memory. Patients will also be complete assessments pre, during and post the intervention to assess and monitor changes to their symptoms.
  Interventions: Other: Narrative Exposure Therapy (NET)

INTERVENTIONS:
Other: Narrative Exposure Therapy (NET) — NET always begins with a face-to-face personal interview between the patient and the therapist to carefully assess life events using checklists, followed by an interview about trauma reactions and a thorough psychoeducation about the findings and suggested procedure of NET. In another session, he arousing and meaningful specific events from birth to present are symbolized in their valence in an autobiographical timeline (or 'lifeline'). The patient is then encouraged to share their life story, focusing on adverse and emotionally charged experiences, which are explored in depth using 'Narrative Exposure', and those are reviewed in the subsequent session.

SUMMARY:
The goal of this interventional study is to evaluate the feasibility of Narrative Exposure Therapy (NET) for people experiencing psychosis. The secondary goal of this study is to evaluate the potential impact of NET in reducing symptoms of psychosis and post-traumatic stress. Participants will be patients accessing local NHS mental health services who are between the age of 18 to 65 years-old who have been diagnosed with a psychotic disorder and have a history of trauma. The main questions the study aims to answer are:

Is NET feasible to deliver to people experiencing psychosis

Can NET impact symptoms of psychosis in people experiencing psychosis?

Can NET impact symptoms posttraumatic stress in people experiencing psychosis?

Can NET impact symptoms of depression, anxiety and stress in people experiencing psychosis?

Participants will be asked to:

Undertake the NET intervention with a trained NET therapist (the number of sessions will be decided based on the need of the participant)

Complete a questionnaire to assess the traumas they have experienced over the course of their life (called the 'Trauma and Life Events' Scale)

Complete a weekly interview to assess their symptoms of psychosis (called the 'Simplified Negative and Positive Symptoms Interview')

Complete weekly measures to assess symptoms of post-traumatic stress (called the 'International Trauma Questionnaire')

Complete weekly measures to assess symptoms of depression, anxiety and stress (using the Depression, Anxiety and Stress 21 item Scale [DASS-21])

Complete a follow-up interview to discuss their personal experience of the NET intervention)

ELIGIBILITY:
Inclusion Criteria: For the purposes of this study the term 'psychosis' covers a range of conditions recognised in standard diagnostic systems such as the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5; APA, 2013) and the International Classification of Diseases - Eleventh Revision (ICD-11; WHO, 2018). Examples include, but are not limited to:

* Schizophrenia Spectrum and Other Psychotic Disorders
* Schizophrenia
* Schizoaffective Disorder
* Brief Psychotic Disorder
* Delusional Disorder
* Substance/Medication-Induced Psychotic Disorder
* Postpartum (Postnatal) Psychosis

Individuals will be eligible to take part in the study if they meet all of the following:

* Age - between 18 and 65 years old.
* Language - able to speak and understand English well enough to take part in the research activities.
* Diagnosis - have a psychosis-related diagnosis as defined above.
* Trauma history - have experienced more than one traumatic event in their lifetime. A traumatic event means something that was deeply distressing, frightening, or life-threatening, such as abuse, assault, serious accident, disaster, or war.
* Current care - are under the care of a Local Mental Health Team (LMHT) within Nottinghamshire Healthcare NHS Foundation Trust and on the Care Programme Approach (CPA) pathway. CPA is an NHS care plan for people with complex mental health needs, setting out the support they will receive and who will provide it.
* Mobility - can travel independently to an NHS clinic or can be supported to attend.
* Consent - able to understand the study information and give informed consent to take part (in line with the Mental Capacity Act, 2005).

Exclusion Criteria: People will not be able to take part in the study if any of the following apply

* Recent change in antipsychotic medication - If the person has recently started, stopped, or changed their antipsychotic medication. This is because there are no specific medical tests ("biomarkers") to predict how someone will respond to a new medication, and the effects can vary greatly between individuals. The first few weeks after a medication change can be a time of increased risk for worsening symptoms or relapse. Research also shows that stopping and starting medication can temporarily affect thinking skills such as memory and attention.

Recent serious mental health crisis -

If the person has experienced a significant adverse event within the last three months, such as:

* A suicide attempt
* A hospital admission for mental health reasons This is because there is currently little research on how trauma-focused therapy affects people with severe mental illness who have recently been suicidal, and starting therapy too soon after a crisis may not be safe.

Currently receiving another structured psychological therapy - For example, Cognitive Behavioural Therapy (CBT) or another regular talking therapy programme. This is to ensure that the results of the study reflect the effects of Narrative Exposure Therapy (NET) alone, without being influenced by another therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Change Interview | The Change Interview will be conducted at the follow-up phase of study which will occur 4 weeks within the final NET session.
  A change interview is a semi-structured interview designed to explore participants' experiences of therapy, its feasibility, acceptability, and perceived effects. It covers general wellbeing, views on specific NET components (psychoeducation, lifeline, questionnaires, session length), and reflections on discussing traumatic memories. Participants are asked about any changes they noticed, the importance of these changes, whether they attribute them to therapy or other factors, and what aspects were helpful or unhelpful. The interview also explores challenges, unexpected experiences, and the significance of specific traumas or positive memories (flowers) discussed in therapy, as well as differences observed between initial and later lifeline sessions.

SECONDARY OUTCOMES:
PANSS-6 | From baseline to the end of follow up which occurs within 4 weeks of the final NET session.
  The PANSS-6 is an abbreviated, clinician-rated version of the 30-item Positive and Negative Syndrome Scale, focused on three core positive symptoms (Delusions - P1, Conceptual Disorganization - P2, Hallucinatory Behavior - P3) and three negative symptoms (Blunted Affect - N1, Passive/Apathetic Social Withdrawal - N4, Lack of Spontaneity and Flow of Conversation - N6). It's psychometrically scalable and sensitive to symptom changes, with accuracy comparable to the full PANSS-30 for assessing severity, remission, and treatment response.
  The PANSS-6 is rated using information collected from the Simplified Negative and Positive Symptoms Interview (SNAPSI) which is a brief semi-structured interview designed to gather information needed to rate the PANSS-6. Clinicians administer the SNAPSI, following its structured probes for each of the six symptom domains, then assign ratings on the 7-point PANSS-6 scale (1 = absent to 7 = extreme) using detailed anchor criteria.
International Trauma Questionnaire (ITQ) | From baseline to the end of follow up which occurs within 4 weeks of the final NET session.
  The International Trauma Questionnaire (ITQ) is a brief, self-report tool aligned with ICD-11, designed to assess both PTSD and Complex PTSD (CPTSD) via 18 items-measuring three core PTSD domains (re-experiencing in the present, avoidance, and sense of current threat), three Disturbances in Self-Organization (DSO) domains (affective dysregulation, negative self-concept, interpersonal difficulties), plus functional impairment for each set of symptoms. Respondents first identify "the experience that troubles you the most" and answer items about symptoms and functioning, rating each from 0 ("not at all") to 4 ("extremely").
DASS-21 (Depression, Anxiety, and Stress Scale) | From baseline to the end of follow up which occurs within 4 weeks of the final NET session.
  The DASS-21 (Depression Anxiety Stress Scales - 21 items) is a short, self-report questionnaire designed to measure the negative emotional states of depression, anxiety, and stress.
  It contains 21 items (7 per subscale).
  Respondents rate how much each statement applied to them over the past week on a 4-point scale (0 = did not apply to me at all, 3 = applied to me very much/most of the time).
  Scores for each subscale (depression, anxiety, stress) are summed and then multiplied by 2 to make them comparable with the longer DASS-42 version.
  It is not a diagnostic tool, but it provides an indication of the severity of symptoms in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schroder, PhD, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: Undecided